CLINICAL TRIAL: NCT04530110
Title: A Multicenter, Open-Label Study Evaluating the Long-Term Safety, Tolerability, and Efficacy of Monthly Subcutaneous Administration of Fremanezumab for the Preventive Treatment of Episodic and Chronic Migraine in Pediatric Patients 6 to 17 Years of Age
Brief Title: A Study to Test if Fremanezumab is Effective in Preventing Migraine in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV48125-CNS-30084; 2019-002056-16 (EudraCT Number); 2024-512837-34-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: episodic migraine; chronic migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fremanezumab (Experimental): The dose of Fremanezumab to be administered will be confirmed or adjusted, as appropriate, based on the participant's weight every 3 months.
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Fremanezumab — Participants weighing ≥ threshold will receive Dose A subcutaneously monthly.
  Participants weighing < threshold will receive Dose B subcutaneously monthly.
  Subcutaneously monthly, confirmed or adjusted, as appropriate, based on the participant's weight every 3 months.

SUMMARY:
The primary objective of the study is to evaluate the long-term safety and tolerability of subcutaneous fremanezumab in the preventive treatment of migraine in pediatric participants 6 to 17 years of age (inclusive at enrollment in the pivotal study).

Secondary objectives are to evaluate the efficacy of subcutaneous fremanezumab in pediatric participants with migraine and to evaluate the immunogenicity of fremanezumab and the impact of ADAs on clinical outcomes in pediatric participants exposed to fremanezumab.

The total duration of the study is planned to be up to 84 months.

DETAILED DESCRIPTION:
The study population will be composed of 3 subgroups of participants as follows:

* Participants rolling over from the pivotal Phase 3 pediatric efficacy studies (Studies TV48125-CNS-30082 and TV48125-CNS-30083)
* Participants rolling over from the Phase 1 pediatric pharmacokinetic study (Study TV48125-CNS-10141)
* Participants rolling over from the pivotal Phase 3 pediatric efficacy studies (Studies TV48125-CNS-30082 and TV48125-CNS-30083) for safety follow-up and antidrug antibody (ADA) evaluation only

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Participants Rolling Over from the Pivotal Efficacy Studies (TV48125-CNS-30082 or TV48125-CNS-30083):

* Participants have completed the pivotal efficacy study and, in the opinion of the Investigator or the Sponsor, are able to complete the study in a safe and compliant way.
* Participants may continue with a stable dose/regimen of the preventive medication they were taking during the pivotal efficacy studies.
* The participant continues to meet appropriate criteria carried forward from the pivotal efficacy study/
* The participant has received all recommended age-appropriate vaccines according to local standard of care and schedule.
* The participant weighs at least 17.0 kg on the day of study enrollment.

NOTE: Additional criteria apply; please contact the investigator for more information.

Inclusion Criteria for Participants Rolling Over from the Phase 1 Pediatric Pharmacokinetic Study (Study TV48125-CNS-10141):

* The participant/caregiver has demonstrated compliance with the electronic headache diary during the 28-day baseline period by entry of headache data on a minimum of 21 out of 28 days (approximately 75% diary compliance).
* The participant has received all recommended age-appropriate vaccines according to local standard of care and schedule.
* The participant weighs at least 17.0 kg on the day of study enrollment.
* The participant has a body mass index ranging from the 5th to 120% of the 95th percentile, inclusive, on the day of study enrollment.
* Not using preventive medications or using no more than 2 preventive medications for migraine or other medical condition, as long as the dose and regimen have been stable for at least 2 months prior to screening (visit 1).

NOTE: Additional criteria apply; please contact the investigator for more information.

Inclusion Criteria for Participants Rolling Over from the Pivotal Efficacy Studies (TV48125-CNS-30082 and TV48125-CNS-30083) for Safety and antidrug antibody (ADA) Assessment Only:

• Participants may be included in this study if they sign and date the informed consent document or upon consent of a parent or guardian, if the participant is younger than the age of consent, accompanied by assent of the participant.

Exclusion Criteria:

Exclusion Criteria for Participants Rolling Over from the Pivotal Efficacy Studies (TV48125-CNS-30082 or TV48125-CNS-30083):

* In the judgment of the investigator, the participant has a clinically significant abnormal finding on study entry, including hematology, blood chemistry, coagulation tests, or urinalysis values/findings (abnormal tests may be repeated for confirmation).
* The participant has a current history of a clinically significant psychiatric condition, at the discretion of the investigator. Any prior history of a suicide attempt, or a history of suicidal ideation with a specific plan within the past 2 years, must be excluded.
* The participant has an ongoing infection or a known history of human immunodeficiency virus infection, tuberculosis, Lyme disease, or chronic hepatitis B or C, or a known active infection of coronavirus disease 2019 (COVID-19).
* The participant has a history of hypersensitivity reactions to injected proteins, including mAbs, or a history of Stevens-Johnson Syndrome or toxic epidermal necrolysis syndrome, or the participant is concomitantly using lamotrigine.
* The participant received a live attenuated vaccine (eg, intranasal flu vaccine, and measles, mumps, and rubella vaccine) within the 12-week period prior to screening. Note: If a medical need arises during the study, the participant may receive a live attenuated vaccine.
* The participant is pregnant or nursing.
* In the judgment of the investigator, the participant has an abnormal finding on the baseline 12-lead ECG considered clinically significant.
* The participant has a current or past medical history of hemiplegic migraine.

NOTE: Additional criteria apply; please contact the investigator for more information.

Exclusion Criteria for Participants Rolling Over from the Phase 1 Pharmacokinetic Study (TV48125-CNS-10141):

* The participant has any clinically significant cardiovascular (including congenital cardiac anomalies or thromboembolic events), endocrine, gastrointestinal, genitourinary, hematologic, hepatic, immunologic, neurologic, ophthalmic, pulmonary, renal disease, or complications of an infection, at the discretion of the investigator.
* The participant has a current history of a clinically significant psychiatric condition, any prior history of a suicide attempt, or a history of suicidal ideation with a specific plan within the past 2 years, at the discretion of the investigator.
* The participant has an ongoing infection or a known history of human immunodeficiency virus infection, tuberculosis, Lyme disease, or chronic hepatitis B or C, or a known active infection of coronavirus disease 2019 (COVID-19).
* The participant has a history of hypersensitivity reactions to injected proteins, including mAbs, or a history of Stevens-Johnson Syndrome or toxic epidermal necrolysis syndrome, or the participant is concomitantly using lamotrigine.
* The participant received a live attenuated vaccine (eg, intranasal flu vaccine, and measles, mumps, and rubella vaccine) within the 12-week period prior to screening. Note: If a medical need arises during the study, the participant may receive a live attenuated vaccine.
* The participant is pregnant or nursing.
* In the judgment of the investigator, the participant has an abnormal finding on the baseline 12-lead ECG considered clinically significant.
* The participant has a current or past medical history of hemiplegic migraine.

NOTE: Additional criteria apply; please contact the investigator for more information.

Exclusion Criteria for Participants Rolling Over from the Pivotal Efficacy Studies (TV48125-CNS-30082 and TV48125-CNS-30083) for Safety and antidrug antibody (ADA) Assessment Only: Not Applicable

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 506 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Day 1 - Day 393
  including local injection site reaction/pain
Incidence of participants with clinically significant changes in laboratory values | Day 1 - Day 253
Incidence of abnormal standard 12-lead electrocardiogram (ECG) findings | Day 1 - Day 253
Incidence of abnormal vital signs | Day 1 - Day 253
  (systolic and diastolic blood pressure, pulse, temperature, and respiratory rate), height, and weight measurements
Incidence of abnormal physical examination findings | Day 1- Day 393
Yes/No suicidality ideation | Day 1 - Day 393
  Columbia-Suicide Severity Rating Scale (C-SSRS) The C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. Scale range: Yes or No response to 10 questions, with minimum to maximum range of 0 to 10. Lower score represents better outcomes.

SECONDARY OUTCOMES:
Mean change in the number of headache days of at least moderate severity | Day 1 - Day 253
Mean change in the number of migraine days | Day 1 - Day 253
Proportion of participants reaching at least 50% reduction in the number of migraine days | Day 1 - Day 253
Proportion of participants reaching at least 50% reduction in the number of headache days of at least moderate severity | Day 1 - Day 253
Mean change in the number of days of use of any acute headache medications | Day 1 - Day 253
Mean change in the PedMIDAS questionnaire score | Day 1 - Day 393
  The Pediatric Migraine Disability Assessment (PedMIDAS) is used to assess migraine disability across multiple domains of functioning including school, home, social, and recreational. The measure consists of 6 items measuring the number of days in which activities were missed as a result of headache/migraine. The measure yields a total score by summing items. Total scores correspond to one of four "disability grades:" 0-10 = little to no disability, 11-30 = mild disability, 31-50 = moderate disability, and >50 = severe disability.
Proportion of participants developing antidrug antibodies (ADAs) throughout the study | Day 1 - Day 393
  The impact of ADAs on safety and efficacy will be analyzed if the number of ADA-positive participants allows.

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (70):
- United States (32):
  - Teva Investigational Site 14319, Aurora, Colorado
  - Teva Investigational Site 14368, Colorado Springs, Colorado
  - Teva Investigational Site 14244, Jacksonville, Florida
  - Teva Investigational Site 14325, Miami, Florida
  - Teva Investigational Site 14250, West Palm Beach, Florida
  - Teva Investigational Site 14255, West Palm Beach, Florida
  - Teva Investigational Site 14243, Atlanta, Georgia
  - Teva Investigational Site 14258, Savannah, Georgia
  - Teva Investigational Site 14263, Hoffman Estates, Illinois
  - Teva Investigational Site 14245, Wichita, Kansas
  - Teva Investigational Site 14327, Louisville, Kentucky
  - Teva Investigational Site 14360, Covington, Louisiana
  - Teva Investigational Site 14365, Baltimore, Maryland
  - Teva Investigational Site 14246, Waltham, Massachusetts
  - Teva Investigational Site 14251, Ann Arbor, Michigan
  - Teva Investigational Site 14270, Minneapolis, Minnesota
  - Teva Investigational Site 14376, Ridgeland, Mississippi
  - Teva Investigational Site 14256, Bridgeton, Missouri
  - Teva Investigational Site 14371, New Brunswick, New Jersey
  - Teva Investigational Site 14276, Amherst, New York
  - Teva Investigational Site 14377, Durham, North Carolina
  - Teva Investigational Site 14248, Raleigh, North Carolina
  - Teva Investigational Site 14264, Cincinnati, Ohio
  - Teva Investigational Site 14257, Oklahoma City, Oklahoma
  - Teva Investigational Site 14363, Tulsa, Oklahoma
  - Teva Investigational Site 14364, Philadelphia, Pennsylvania
  - Teva Investigational Site 14374, Bristol, Tennessee
  - Teva Investigational Site 14252, Austin, Texas
  - Teva Investigational Site 14273, Austin, Texas
  - Teva Investigational Site 14367, Dallas, Texas
  - Teva Investigational Site 14375, Salt Lake City, Utah
  - Teva Investigational Site 14323, Norfolk, Virginia
- Canada (3):
  - Teva Investigational Site 11182, Ottawa, Ontario
  - Teva Investigational Site 11179, Ottawa, Ontario
  - Teva Investigational Site 11181, Montreal, Quebec
- Finland (4):
  - Teva Investigational Site 40053, Helsinki
  - Teva Investigational Site 40049, Kuopio
  - Teva Investigational Site 40054, Oulu
  - Teva Investigational Site 40052, Tampere
- Germany (3):
  - Teva Investigational Site 32728, Bad Homburg
  - Teva Investigational Site 32729, Berlin
  - Teva Investigational Site 32726, Leipzig
- Israel (7):
  - Teva Investigational Site 80170, Be’er Ya‘aqov
  - Teva Investigational Site 80166, Haifa
  - Teva Investigational Site 80168, Holon
  - Teva Investigational Site 80169, Jerusalem
  - Teva Investigational Site 80167, Ramat Gan
  - Teva Investigational Site 80164, Safed
  - Teva Investigational Site 80165, Tel Aviv
- Italy (7):
  - Teva Investigational Site 30230, Florence
  - Teva Investigational Site 30239, Milan
  - Teva Investigational Site 30228, Milan
  - Teva Investigational Site 30226, Milan
  - Teva Investigational Site 30238, Padua
  - Teva Investigational Site 30227, Pavia
  - Teva Investigational Site 30225, Rome
- Netherlands (3):
  - Teva Investigational Site 38138, Doetinchem
  - Teva Investigational Site 38135, Nijmegen
  - Teva Investigational Site 38136, Rotterdam
- Poland (8):
  - Teva Investigational Site 53441, Gdansk
  - Teva Investigational Site 53437, Kielce
  - Teva Investigational Site 53443, Krakow
  - Teva Investigational Site 53452, Krakow
  - Teva Investigational Site 53440, Lublin
  - Teva Investigational Site 53439, Poznan
  - Teva Investigational Site 53451, Poznan
  - Teva Investigational Site 53442, Szczecin
- Spain (3):
  - Teva Investigational Site 31271, Barcelona
  - Teva Investigational Site 31270, Valencia
  - Teva Investigational Site 31265, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.